CLINICAL TRIAL: NCT03936647
Title: The RISE Trial: A Randomized Trial on Intra-Saccular Endobridge Devices
Acronym: RISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-8330
Record Dates: First submitted 2019-04-17; First posted 2019-05-03 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Intracranial Aneurysm; Brain Aneurysm; Unruptured Cerebral Aneurysm; Ruptured Cerebral Aneurysm; Cerebral Aneurysm
Keywords: intracranial aneurysm; cerebral aneurysm; brain aneurysm; unruptured cerebral aneurysm; ruptured cerebral aneurysm; WEB embolization device; embolization
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Intervention Model Description: Standard best conventional treatment option (surgical or endovascular) vs WEB embolization device
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard conventional treatment (surgical or endovascular) (Active Comparator): Treatment may include the most appropriate amongst surgical clipping, simple coiling, high-porosity stenting with or without coiling, and intra-arterial flow diversion with or without coiling, which will be predetermined by the treating physician prior to randomization.
  Interventions: Procedure: surgical clipping, simple coiling, high-porosity stenting with/ without coiling, intra-arterial flow diversion with/ without coiling
- WEB embolization device (Experimental): Endovascular treatment with WEB, including standard management of thrombo-embolic risk
  Interventions: Device: WEB embolization device

INTERVENTIONS:
Procedure: surgical clipping, simple coiling, high-porosity stenting with/ without coiling, intra-arterial flow diversion with/ without coiling — Treatment may include the most appropriate amongst surgical clipping, simple coiling, high-porosity stenting with or without coiling, and intra-arterial flow diversion with or without coiling, which will be predetermined by the treating physician prior to randomization.
  Arms: Standard conventional treatment (surgical or endovascular)
Device: WEB embolization device — WEB embolization device
  Arms: WEB embolization device

SUMMARY:
Intracranial bifurcation aneurysms are commonly repaired with surgical and with endovascular techniques. Wide-necked bifurcation aneurysms (WNBA) are a difficult subset of aneurysms to successfully repair endovascularly, and a number of treatment adjuncts have been designed. One particularly promising innovation is the WEB (Woven EndoBridge), which permits placement of an intra-saccular flow diverting mesh across the aneurysm neck, but which does not require anti-platelet agent therapy. Currently, which treatment option leads to the best outcome for patients with WNBA remains unknown. There is a need to offer treatment with the WEB within the context of a randomized care trial, to patients currently presenting with aneurysms thought to be suitable for the WEB.

ELIGIBILITY:
Inclusion Criteria:

* patient with an intracranial aneurysm in whom WEB is considered an appropriate therapeutic option by the participating clinician
* aneurysm of maximum diameter of 4-11 mm
* may include (but are not restricted to) saccular bifurcation aneurysms of the middle cerebral artery, basilar bifurcation, carotid terminus, or anterior communicating artery aneurysms
* Recurring, persistent aneurysm after previous treatment can be included so long as the treating physician judges the aneurysm morphology to be appropriate.
* Ruptured aneurysms with WFNS ≤ 3

Exclusion Criteria:

* Absolute contraindication to surgery, endovascular treatment or anesthesia
* Patients unable to give informed consent
* diameter of the aneurysm ≤ 4 mm but ≥ 11 mm
* Ruptured aneurysms with WFNS 4 or 5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-07-18 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with imaging showing that index aneurysm has reached complete or near occlusion | 1 year from procedure
  complete or near complete occlusion of the aneurysm
Number of patients with a modified Rankin Score (mRS) below or equal to 2 | 1 year from procedure
  mRS ≤2 from evaluation (questionnaire) at follow-up visits throughout study. Grading score is to be assessed as such: Grade 0 No symptoms at all. Grade 1 No significant disability despite symptoms; able to carry out all usual duties and activities Grade 2 Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance Grade 3 Moderate disability; requiring some help, but able to walk without assistance Grade 4 Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance Grade 5 Severe disability; bedridden, incontinent and requiring constant nursing care and attention Grade 6 Dead

SECONDARY OUTCOMES:
Number of participants with an interim modified Rankin Scale (mRS) below or equal to 2 | within 1 week post-procedure, 1-3 months, and 12 months post-treatment
  mRS ≤2 from evaluation (questionnaire) at discharge and follow-up visits throughout study. Grading score is to be assessed as such: Grade 0 No symptoms at all. Grade 1 No significant disability despite symptoms; able to carry out all usual duties and activities Grade 2 Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance Grade 3 Moderate disability; requiring some help, but able to walk without assistance Grade 4 Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance Grade 5 Severe disability; bedridden, incontinent and requiring constant nursing care and attention Grade 6 Dead
Number of successful deployment of WEB device, coils or successful microsurgical, clipping, along with judgement of patency of parent arteries using imaging (depending on treatment received) | within 1 hour from procedure
  Successful WEB deployment / aneurysm clipping / aneurysm coiling
Number of incidences of successful or unsuccesful patency of parent arteries using imaging | within 1 hour from procedure
  Analysis of imaging to judge the patency of the parent arteries
Number of peri-operative complications | ≥5 days
  Peri-operative complications (such as ischemic strokes and intracranial hemorrhages)
Number of aneurysm re-occurrences, (re-)rupture, or incomplete occlusion based on angiographic imaging | 12 +/- 2 months
  Angiographic outcome (invasive or non-invasive imaging) results
Hospitalization time | up to first post-procedure visit (around 1 month)
  Hospital stay (number of days)
Incidence of discharge destination by type | up to first post-procedure visit (around 1 month)
  Discharge disposition (home; other hospital; rehabilitation facility; death)
Number of participants with stroke, neurological symptom or sign | within 12 +/- 2 months
  Any new stroke, neurological symptom or sign
Number of index aneurysms necessitating or having received retreatment due to re-occurence | Within 12 +/- 2 months
  Re-treatment of the index aneurysm as judged by imaging and interventionists neurosurgeons due to incomplete occlusion or hemorrhage

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - University of Alberta Hospital, Edmonton, Alberta
  - University of Manitoba Hospital, Winnipeg, Manitoba
  - Hamilton Health Sciences - McMaster University, Hamilton, Ontario
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No